CLINICAL TRIAL: NCT03561051
Title: The Pre-hospital Evaluation of Sensitive Troponin (PRESTO) Study
Status: Active, not recruiting | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Abbott Point of Care (Industry); LumiraDx (Industry); Roche Diagnostics GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: B00041; 223790 (Other: IRAS Project ID)
Record Dates: First submitted 2018-06-06; First posted 2018-06-19 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Chest Pain; Acute Coronary Syndrome; Heart Attack
Keywords: T-MACS; Pre-hospital environment
MeSH Terms: conditions — Chest Pain; Acute Coronary Syndrome; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to assess whether a decision aid that is currently used in hospitals across Greater Manchester to determine how likely it is that a patient has a serious heart problem is still accurate in the pre-hospital environment.

DETAILED DESCRIPTION:
The Investigators will aim to recruit up to 700 participants, aged 18-100, who call 999 with a complaint of chest pain and are subsequently attended by the ambulance service. A blood sample will be taken in the ambulance as well as information about the participant's symptoms, past medical history, physical examination findings and heart tracing findings. The participant will then be transferred to hospital, where another blood sample will be taken. Both of these blood samples will be analysed at a later date for the cardiac marker, troponin.

Participants will then be followed up after 30 days via screening of their clinical records and contacting their GP. The investigators will gather information on the participant's initial admission to hospital, as well as any further hospital admissions and investigations that have occurred within the 30 days since this admission. The information collected will include data on serial cardiac marker testing; other laboratory analyses; length of stay; all imaging investigations and procedures; and details of any haemorrhagic complications.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years)
* Called 999 for an emergency ambulance because they have experienced pain, discomfort or pressure in the chest, epigastrium, neck, jaw or upper limb without an apparent non-cardiac source
* Treating paramedic suspects these symptoms may be caused by acute coronary syndromes.

Exclusion Criteria:

* Patients with unequivocal evidence of ST elevation myocardial infarction who are being immediately transferred for primary percutaneous coronary intervention
* Patients in whom an alternative diagnosis (other than acute coronary syndromes) is suspected, which would necessitate transfer to hospital
* Patients who have not experienced symptoms in the previous 24 hours
* Patients who lack the capacity to provide written informed consent, either because they lack the mental capacity to provide written informed consent or because effective communication is not possible (e.g. non-English speakers in the absence of adequate translation services)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will recruit patients who have called 999 with a complaint of pain, discomfort or pressure in the chest, who are then attended by an ambulance.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2018-10-16 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of acute myocardial infarction | 30 days

SECONDARY OUTCOMES:
Incident major adverse cardiac events | 30 days
Prevalent acute myocardial infarction | 30 days
Final diagnosis of participant | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Richard Body, Principal Investigator — Manchester University NHS Foundation Trust
Locations (13):
- United Kingdom (13):
  - Bolton NHS Foundation Trust, Bolton
  - North West Ambulance Service NHS Trust, Bolton
  - North Bristol NHS Trust, Bristol
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - West Midlands Ambulance Service NHS Foundation Trust, Dudley
  - Royal Devon and Exeter NHS Foundation Trust, Exeter
  - South Western Ambulance Service NHS Foundation Trust, Exeter
  - Manchester University NHS Foundation Trust, Manchester
  - Plymouth Hospitals NHS Trust, Plymouth
  - Salford Royal NHS Foundation Trust, Salford
  - Taunton and Somerset NHS Foundation Trust, Taunton
  - South Warwickshire NHS Foundation Trust, Warwick
  - Wrightington, Wigan and Leigh NHS Foundation Trust, Wigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gilman J, Alghamdi A, Hann M, Carlton E, Cooper JG, Cook E, Siriwardena AN, Phillips J, Thompson A, Bell S, Kirby K, Rosser A, Body R. Diagnostic Accuracy of a Novel Point of Care High-Sensitivity Troponin Assay in the Prehospital Environment. Acad Emerg Med. 2026 Jan;33(1):e70213. doi: 10.1111/acem.70213. PMID 41528153
- [Derived] Alghamdi A, Hann M, Carlton E, Cooper JG, Cook E, Foulkes A, Siriwardena AN, Phillips J, Thompson A, Bell S, Kirby K, Rosser A, Body R. Diagnostic Accuracy of Clinical Pathways for Suspected Acute Myocardial Infarction in the Out-of-Hospital Environment. Ann Emerg Med. 2023 Oct;82(4):439-448. doi: 10.1016/j.annemergmed.2023.04.010. Epub 2023 Jun 10. PMID 37306636
- [Derived] Alghamdi A, Cook E, Carlton E, Siriwardena A, Hann M, Thompson A, Foulkes A, Phillips J, Cooper J, Bell S, Kirby K, Rosser A, Body R. PRe-hospital Evaluation of Sensitive TrOponin (PRESTO) Study: multicentre prospective diagnostic accuracy study protocol. BMJ Open. 2019 Oct 28;9(10):e032834. doi: 10.1136/bmjopen-2019-032834. PMID 31662404